CLINICAL TRIAL: NCT03513926
Title: Molecular Profile of Cardiovascular Risk in Obstructive Sleep Apnea Patients: Personalized Predictive Model.
Status: Completed | Type: Observational
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Principal Investigator, Ferran Barbe, Medical Doctor, Sociedad Española de Neumología y Cirugía Torácica
Other Study IDs: PI14/01266
Record Dates: First submitted 2017-05-04; First posted 2018-05-02 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Obstructive Sleep Apnea; Hypertension; Cardiovascular Diseases
Keywords: miRNA; Cardiovascular Risk; CPAP; Obstructive Sleep Apnea; Hypertension; Molecular profile
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension; Cardiovascular Diseases | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Serum, Plasma and buffy coat
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (4):
- Non-OSA group: Patients with out sleep apnea.
- OSA group: Patients with OSA, without cardiovascular comorbidities who could be treated with Continuous Positive Airway Pressure
  Interventions: Device: Continuous Positive Airway Pressure
- OSA with hypertension group: Patients with OSA, with hypertension who could be treated with Continuous Positive Airway Pressure
  Interventions: Device: Continuous Positive Airway Pressure
- OSA with CVE group: Patients with OSA, with a previous ictus or stroke who could be treated with Continuous Positive Airway Pressure
  Interventions: Device: Continuous Positive Airway Pressure

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — Continuous Positive Airway Pressure
  Other Names: CPAP
  Groups: OSA group; OSA with CVE group; OSA with hypertension group

SUMMARY:
Evaluation of anthropometric, clinical and biological profile in four groups that represents transversely the natural history of Obstructive Sleep Apnea (OSA) and its associated cardiovascular comorbidities: non-OSA, OSA without hypertension, OSA and with hypertension and OSA with a cardiovascular event (CVE).

DETAILED DESCRIPTION:
Aims: The main objective of the study is to determine the risk profile associated with the development of cardiovascular (CV) disease in patients with OSA. To do this, by using genomic analysis tools, transcriptome and the analysis of protein markers are established the following objectives: 1) to determine differences in phenotypic profile (anthropometric, clinical, analytical and biological variables) from different populations: non-hypertensive patient with OSA, OSA hypertensive patient, OSA hypertensive patient who has developed a CV event and healthy subject. These four populations represent transversely the natural history of OSA. In this way the phenotype of the OSA patient and its relationship with risk of developing of CV disease will be defined. 2) To define the changes produced in these profiles after effective treatment with continuous positive airway pressure (CPAP). This approach allows to evaluate the different pathogenic pathways related to CV risk in patients with OSA. 3) To define a predictive model of cardiovascular risk and response to CPAP treatment, in patients with OSA. 4) To phenotype and define the different and segregated clusters of OSA patients whose recognition may improve prognostic predictions and guide therapeutic strategies Methodology: For ethical reasons a longitudinal study cannot be carried out to know history natural the disease (can not leave without treatment patients with OSA long term). We propose a transversal study in which will be include four populations that representing transversally the natural history of OSA (non-OSA individuals, non-hypertensive OSA patients, OSA patients with hypertension and hypertensive OSA patients who have developed a CV event). All the patients will be performed a general analysis, lipid profile and polysomnography. The expression profile of microRNAs associated with cardiovascular risk will be assessed in addition to the gene expression profile associated with arterial hypertension. The measurements are made at baseline and 6 months after effective treatment with CPAP. This methodological approach will contribute in the identification of OSA phenotype which could develop cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with suspected OSA that attend to Sleep Unit of Hospital Arnau de Vilanova- Santa Maria de Lleida.
* 18-60 years old

Exclusion Criteria:

* Any chronic disease (malignancy, renal insufficiency (glomerular filtration rate <30 ml / min), severe chronic obstructive pulmonary disease, chronic depression and other chronic diseases very limiting),
* Any sleep disorder previously diagnosed: narcolepsy, insomnia, chronic lack of sleep, regular use of hypnotic or sedative drugs and restless leg syndrome
* Any genetic abnormality or disease
* Any medical, social or geographical factors which may endanger patient compliance. (For example, consumption of alcohol (more than 80 g / day in men and 60 g / day in women), disorientation, or a history of default).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Suspected OSA patients attending consecutively to the Sleep Unit of the University Hospital Arnau de Vilanova- Santa María de Lleida are included.
Sampling Method: Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Modeling the cardiovascular (CV) disease risk in patients with obstructive sleep apnea (OSA) through the analysis of the number and specific biomarkers. | Baseline
  Anthropometric, clinical, analytical and biological variables characterization from different populations:non-OSA, OSA without hypertension, OSA with hypertension and OSA with a CV event. The evaluation of these variables will permit the characterization of the profile associated with CV disease in patients with OSA.

SECONDARY OUTCOMES:
Modeling the effect of the treatment with continuous positive airway pressure (CPAP) in patients with OSA with and without cardiovascular disease, through the analysis of the number and specific biomarkers. | After 6 months of follow-up
  Anthropometric, clinical, analytical and biological variables characterization from different populations:non-OSA, OSA without hypertension, OSA with hypertension and OSA with a CV event. The evaluation of these variables changes after CPAP treatment will allow to characterize the effect of this treatment in biomarker related with CV disease
Predictive model of cardiovascular risk | After 6 months of follow-up
  Define a predictive model of cardiovascular risk and response to CPAP treatment, in patients with OSA.

CONTACTS AND LOCATIONS:
Overall Officials: Ferran Barbé, MD, Principal Investigator — Sociedad Española de Neumología y Cirugía Torácica; Manuel Sanchez-de-la-Torre, PhD, Principal Investigator — Consorcio Centro de Investigación Biomédica en Red (CIBER)
Locations (1):
- Hospital Universitario Santa Maria de Lleida, Lleida, Spain

IPD SHARING:
Plan to Share IPD: Undecided